CLINICAL TRIAL: NCT03244410
Title: Initial Lymphocyte Counts Predictive Value in Immune Thrombocytopenic Purpura
Brief Title: Lymphocyte Counts in Immune Thrombocytopenic Purpura
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dolagy nabil naguib, principle investigator, Assiut University
Other Study IDs: LCITP
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- immune thrombocytopenic purpura: immune thrombocytopenic purpura an acquired autoimmune disorder characterized by increased platelet destruction and decreased platelet number we used complete blood picture
  Interventions: Diagnostic Test: complete blood picture

INTERVENTIONS:
Diagnostic Test: complete blood picture — complete blood picture

SUMMARY:
* immune thrombocytopenic purpura is an acquired autoimmune disorder characterized by increased platelet destruction and decreased platelet number (cooper N et al 2006)
* recent studies have demonstrated that the pathogenesis of ITP envolves multifactorial autoimmune mechanisms of both humoral and cellular immunity and that acute and chronic forms may represent two distinct immunopathological disorders ( cooper N et al 2006) ( Gern Sheimer T 2009 )

DETAILED DESCRIPTION:
Immune thrombocytopenic purpura is an acquired autoimmune disorder characterized by increased platelet destruction and decreased platelet number ( Cooper N et all 2006) platelet surface membrane proteins become antigenic for unknown reasons, leading to stimulation of the immune system, auto antibodies production and platelet destruction ( Gasbarrini A et all 2000) It is associated with the production of auto antibodies directed against platelet glycoprotein complex 2b/3a and/or 1b/1x , resulting in accelerated destruction of platelets by the reticular endothelial system via the activity of Fcc receptor bearing phagocytic cells ( Provan & Newland et al 2002) Recent studies have demonstrated that the pathogenesis of ITP envolves multifactorial autoimmune mechanisms of both humoral and cellular immunity and that acute and chronic forms may represent two distinct immunopathological disorders ( Cooper N et al 2006) ( Gern Sheimer T 2009)

There are many phases of the disease:

1. Newly diagnosed ITP : for all cases at diagnosis.
2. persistent ITP: for patients with ITP between 3 to 12 months.
3. chronic ITP: for patients with ITP lasting more than one year ( blood journal 2009).

   * Although lymphocytopenia is a commonly reported feature of many chronic autoimmune disorders, differential white cell counts at presentation have seldom been evaluated as predictors for development of chronic ITP ( Deel MD et al 2013) (Ahmed et al 2010)

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cases of primary ITP , adults and children.

Exclusion Criteria:

* Cases of secondary ITP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary immune Thrombocytopenic Purpura
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
lymphocyte count in immune thrombocytopenic purpura | 15 minutes
  intital lymphocyte counts predictive value in immune thrombocytopenic purpura by complete blood picture